CLINICAL TRIAL: NCT00623181
Title: Preference for Fluzone Vaccine Administered Intradermally Versus Intramuscularly in Healthy Adult Subjects 18-49 Years of Age
Brief Title: Study to Determine a Preference for Fluzone Vaccine Given Intradermally (ID) and Intramuscularly (IM) in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FID30
Record Dates: First submitted 2008-02-06; First posted 2008-02-25 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza; Influenza virus
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluzone Intradermal First, Then Fluzone Intramuscular (Experimental)
  Interventions: Biological: Fluzone: Influenza virus vaccine
- Fluzone Intramuscular First, Then Fluzone Intradermal (Experimental)
  Interventions: Biological: Fluzone: Influenza virus vaccine

INTERVENTIONS:
Biological: Fluzone: Influenza virus vaccine — 0.1 mL, Intradermal Right deltoid, 0.5 mL, Intramuscular Left deltoid
  Other Names: Fluzone®
  Arms: Fluzone Intradermal First, Then Fluzone Intramuscular
Biological: Fluzone: Influenza virus vaccine — 0.5 mL, Intramuscular Right deltoid, 0.1 mL, Intradermal Left deltoid
  Other Names: Fluzone®
  Arms: Fluzone Intramuscular First, Then Fluzone Intradermal

SUMMARY:
To describe any degree of preference for the route of administration of Fluzone influenza vaccine, ID versus IM, in healthy adult subjects 18-49 years of age.

To collect safety data, injection site reactions, and systemic reactions, through Day 7 post-vaccination; SAEs through day 28 post-vaccination

DETAILED DESCRIPTION:
The purpose of this clinical trial is to determine, in a relatively small sample of persons 18-49 years of age, if there is a preference trend for a particular route of administration, ID vs IM, when receiving a seasonal influenza vaccine. Uptake of influenza vaccine is disappointingly low in this age group, and there is the perception that aversion to IM injection plays a role in vaccination avoidance. The BD Micro-Injection System to be used in this study may offer a more acceptable alternative to the standard IM injection for influenza immunization and thereby promote wider acceptance of influenza vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject (can have underlying medical condition, as long as they are stable), greater than or equal to 18 to < 50 years of age on the day of inclusion.
* Informed consent form signed.
* Able to attend both scheduled visits and to comply with all trial procedures.
* For a woman of child-bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to vaccination, until at least 4 weeks after vaccination.

Exclusion Criteria:

* Subject currently breast-feeding.
* Participation in another investigational clinical trial in the 4 weeks preceding and during the trial period.
* Hypersensitivity to egg proteins, chicken proteins, or to any of the vaccine components, or history of a life-threatening reaction to the trial vaccine or a vaccine containing any of the same substances.
* Thrombocytopenia or bleeding disorder contraindicating IM vaccination.
* Any other condition which in the opinion of the Investigator would pose a health risk to the subject or interfere with the evaluation of the vaccine.
* Personal history of Guillain-Barre syndrome.
* Current use of alcohol or recreational drugs that in the opinion of the Investigator might interfere with the subject's ability to comply with trial procedures.
* Febrile illness (oral temperature greater than or equal to 99.5 degrees F) on day of inclusion (temporary deferral).
* Influenza vaccination received this season (2007-2008).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur, Inc
Locations (2):
- United States (2):
  - Grove City, Pennsylvania
  - Pittsburgh, Pennsylvania

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated from 25 January 2008 to 11 March 2008 in 1 medical center in the US.
Pre-assignment Details: A total of 110 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Fluzone Intradermal First, Then Fluzone Intramuscular: Participants who received 1 dose of Fluzone Intradermal (ID) in the right deltoid region, followed by Fluzone Intramuscular (IM) in the left deltoid region on Day 0
- Fluzone Intramuscular First, Then Fluzone Intradermal: Participants who received 1 dose of Fluzone Intramuscular in the right deltoid region, followed by Fluzone Intradermal (ID) in the left deltoid region on Day 0
Period: Overall Study
Arm/Group | Fluzone Intradermal First, Then Fluzone Intramuscular | Fluzone Intramuscular First, Then Fluzone Intradermal
Started | 56 | 54
Completed | 56 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone Intradermal First, Then Fluzone Intramuscular | Fluzone Intramuscular First, Then Fluzone Intradermal | Total
Number analyzed (Participants) | 56 | 54 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 54 | 110
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.2 (11.44) | 31.3 (10.58) | 31.27 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 24 | 59
  Male | 21 | 30 | 51
Region of Enrollment [Number; unit: participants]
  United States | 56 | 54 | 110

OUTCOME MEASURES:

1. Primary Outcome: Categorical Summary of Pain or Other Discomfort Immediately After Vaccination and on Days 3 and 7 Post-vaccination
Description: Pain or other discomfort was assessed on a scale of 0 to 10 (None = 0; Hardly Any = 1, 2; Mild = 3, 4; Moderate = 5, 6; Severe = 7, 8; Unbearable = 9, 10) according to route of administration: intradermal (ID) as Group 1 and intramuscular (IM) as Group 2.
  Data for this outcome were combined for responses following a similar type of vaccination route in the entire study population.
Time Frame: Day 0 and up to 7 days post-vaccination
Population: Pain or other discomfort was assessed in the Per-Protocol Population. Data were combined for responses following a similar type of vaccination route.
Measure: Number; unit: Participants
Groups:
- Fluzone Intradermal Vaccine: Responses of participants following the receipt of a dose of Fluzone Intradermal (ID) in the right deltoid region or the left deltoid region on Day 0
- Fluzone Intramuscular Vaccine: Responses of participants following the receipt of a dose of Fluzone Intramuscular (IM) in the right deltoid region or the left deltoid region on Day 0
Arm/Group | Fluzone Intradermal Vaccine | Fluzone Intramuscular Vaccine
Number analyzed (Participants) | 101 | 101
Participants
  Any - Day 0 | 85 | 75
  Severe or Worse - Day 0 | 4 | 2
  Any - Day 3 | 44 | 35
  Severe or Worse - Day 3 | 0 | 0
  Any - Day 7 | 5 | 4
  Severe or Worse - Day 7 | 0 | 0

2. Primary Outcome: Continuous Summary of Pain or Other Discomfort Immediately After Vaccination and on Days 3 and 7 Post-vaccination
Description: Numerical scores were assigned to pain by participants on the preference questionnaire as: None = 0; Hardly Any = 1, 2; Mild = 3, 4; Moderate = 5, 6; Severe = 7, 8; or Unbearable = 9, 10.
  Data for this outcome were combined for responses following a similar type of vaccination route in the entire study population.
Time Frame: Days 0, 3, and 7 after vaccination
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Fluzone Intradermal Vaccine | Fluzone Intramuscular Vaccine
Number analyzed (Participants) | 101 | 101
Scores on a scale
  Day 0 | 2.97 (2.13) | 2.02 (1.90)
  Day 3 | 0.79 (1.23) | 0.68 (1.20)
  Day 7 | 0.08 (0.39) | 0.05 (0.26)

3. Other Pre Specified Outcome: Number of Participants Reporting Any Solicited Injection Site Reactions After Vaccine Injection
Description: Solicited injection site reactions: Pain, Pruritus, Erythema, Swelling, Induration, Ecchymosis.
  Data for this outcome were combined for responses following a similar type of vaccination route in the entire study population.
Time Frame: Days 0 through 7 post-vaccination
Population: Safety parameters were assessed in all enrolled and vaccinated participants, intend-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Fluzone Intradermal Vaccine | Fluzone Intramuscular Vaccine
Number analyzed (Participants) | 110 | 110
Participants
  Any Solicited Injection Site Pain | 70 | 75
  Gr 3 Solicited Injection Site -Pain Incapacitating | 0 | 1
  Any Solicited Injection Site Pruritus | 39 | 12
  Gr 3 Solicited Inj. Siite Pruritus -Incapacitating | 1 | 0
  Any Solicited Injection Site Erythema | 92 | 15
  Grade 3 Solicited Injection Site Erythema (≥ 5 cm) | 11 | 0
  Any Solicited Injection Site Swelling | 68 | 12
  Grade 3 Solicited Injection Site Swelling (≥ 5 cm) | 1 | 0
  Any Solicited Injection Site Induration | 74 | 19
  Gr 3 Solicited Injection Site Induration (≥ 5 cm) | 1 | 0
  Any Solicited Injection Site Ecchymosis | 14 | 7
  Gr 3 Solicited Injection Site Ecchymosis (≥ 5 cm) | 0 | 0

4. Other Pre Specified Outcome: Number of Participants Reporting Solicited Systemic Reactions After Vaccine Injection
Description: Solicited systemic reactions: Fever (temperature); Headache; Malaise; and Myalgia.
  Data for this outcome were based on the first vaccination type, intradermal or intramuscular.
Time Frame: Days 0 through 7 post-vaccination
Population: Safety parameters were assessed in all enrolled and vaccinated subjects, intend-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Fluzone Intradermal First, Then Fluzone Intramuscular | Fluzone Intramuscular First, Then Fluzone Intradermal
Number analyzed (Participants) | 56 | 54
Participants
  Any Solicited Fever | 6 | 3
  Grade 3 Solicited Fever (> 102.2 °F) | 0 | 0
  Any Solicited Headache | 25 | 25
  Gr 3 Solicited Headache -Prevents daily activities | 3 | 1
  Any Solicited Malaise | 18 | 21
  Gr 3 Solicited Malaise (Prevents daily activities) | 4 | 4
  Any Solicited Myalgia | 31 | 26
  Gr 3 Solicited Myalgia (Prevents daily activities) | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the day of vaccination for up to 28 days post-vaccination.
Arm/Group | Fluzone Intradermal First, Then Fluzone Intramuscular | Fluzone Intramuscular First, Then Fluzone Intradermal
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/54
Other Adverse Events (participants affected / at risk) | 92/110 | 75/110
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Fluzone Intradermal First, Then Fluzone Intramuscular (N=110) | Fluzone Intramuscular First, Then Fluzone Intradermal (N=110)
Injection Site Pain (General disorders) | 70 (70) | 75 (75)
Injection Site Pruritus (General disorders) | 39 (39) | 12 (12)
Injection Site Erythema (General disorders) | 92 (92) | 15 (15)
Injection Site Swelling (General disorders) | 68 (68) | 12 (12)
Injection Site Induration (General disorders) | 74 (74) | 19 (19)
Injection Site Ecchymosis (General disorders) | 14 (14) | 7 (7)
Fever (General disorders) | 6/56 (6) | 3/54 (3)
Malaise (General disorders) | 18/56 (18) | 21/54 (21)
Headache (Nervous system disorders) | 25/56 (25) | 25/54 (25)
Myalgia (Musculoskeletal and connective tissue disorders) | 31/56 (31) | 26/54 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.